CLINICAL TRIAL: NCT06654765
Title: Growth and Development of Children With Inborn Errors of Metabolism in Assiut Governorate
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Abd El-mohsen Mahfouz, Assistant lecturer, Assiut University
Other Study IDs: Inborn errors of metabolism
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Inborn Errors of Metabolism
Keywords: Growth; Development; IEM; Assiut
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Assessment of growth and development of children with inborn errors of metabolism in Assiut Governorate

DETAILED DESCRIPTION:
Inborn errors of metabolism (IEM) are diseases resulting in deficient activity of an individual enzyme, structural protein in an intermediate metabolic pathway, present clinically in a wide variety of ways a ranging from non-specific chronic issues such as childhood delay in attaining development milestones, to acute decompensation.

The prevalence of all of inborn errors of metabolism globally is 50.9/100000 live birth, In Egypt the prevalence among clinically suspected children is 7.8%.

A study conducted in Minia Governorate (Egypt) on children less than 18 years included 67 children showed that 65.7% of children were under height. Also a study conducted in upper Egypt on 113 PKU patients showed that global developmental delay 54.9% was the most frequent presentations of PKU children. Parents of children with IEM face many challenges; as the financial burden and perceived restrictions in all aspects of life, discrimination by society in general, and the main challenge is dietary restrictions.

Rationale:

Despite being rare in Egypt, IEM are regarded as a national priority because of the substantial health burden they place on the growth and development of the affected children, which can range from delayed achievement of developmental milestones to acute decompensation and death.

However, there is lack of longitudinal studies in Egypt that focus on how IEM affect physical development and growth, as well as the difficulties parents encounter while caring for their children and following up with them. To our knowledge, no local studies have been conducted in this field before.

ELIGIBILITY:
Inclusion Criteria:

* Under five years old children with confirmed diagnosis of IEM.
* Attending the study settings.

Exclusion Criteria:

* Patients diagnosed since birth with dysmorphic features.
* Patients diagnosed since birth with congenital anomalies.
* Patients with other neurological deficits (e.g. cerebral palsy, convulsions, birth anoxia…..)

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Under five years old children with confirmed diagnosis of IEM who are attending the study settings
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
• To assess weight (in kilograms) of children with IEM in Assiut governorate. | 1 year
  The weight will be measured to the nearest 0.1Kg and the patients in light clothes and bare feet.
  The child weight will be measured and the measurements will be plotted on the Egyptian growth charts of girls and boys for different ages from birth to five years old in order to assess their growth.
• To assess height (in meters) of children with IEM in Assiut governorate. | 1 year
  If the child is less than 2 years old or is unable to stand recumbent length will be measured to the nearest 0.1 cm.
  If the child is aged 2 years or older and able to stand, standing height will be measured to the nearest 0.1 cm.
  The child height will be measured and the measurements will be plotted on the Egyptian growth charts of girls and boys for different ages from birth to five years old in order to assess their growth.
• To assess the body mass index for age (BMI for age in kg/m^2) of children with IEM in Assiut governorate. | 1 year
  Body mass index for age (BMI for age) will be calculated in kg/m^2 and plotted on the Egyptian growth charts of girls and boys for different ages from birth to five years old in order to assess their growth.
To assess development of children with IEM in Assiut governorate using the arabic version of the third edition of the Ages and Stages Questionnaires. | 1 year
  The Arabic version of the third edition of the Ages & Stages Questionnaires (ASQ-3) will be used to identify developmental growth in children from one month to five and a half years .
  it measures development in 5 key domains: communication, gross motor, fine motor, problem solving, and personal-social domain.
  Each response on the questionnaire will be converted to a numerical value (usually equal to 10, occasionally to 5, and not yet to 0) in order to determine the score, then each domain's overall score will be summed. ASQ-3 has three scoring zones and the higher the score the better the child development for each developmental area separately.
• To assess knowledge of the mother regarding the child metabolic disease and dietary recommendations using a questionnaire to be designed. | 1 year
  Knowledge regarding the child inborn metabolic diseases such as disease definition, symptoms necessitate immediate hospital admission, disease complications, dietary requirement and restrictions.
Assessment of mother's practice using a questionnaire to be designed. | 1 year
  Dietary practice, child care, vaccination and follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Sabra Mohamed Ahmed, Prof. Dr, Study Director — Assiut University; Taghreed Abdel-Aziz Mohamed, Prof. Dr, Study Director — Assiut University; Samar Mahfouz, assistant lecturer, Principal Investigator — Assiut University
Locations (1):
- • Genetic counselling center at Al Weladea neighbourhood in Assiut governorate. • Genetics Center at Al-Iman General Hospital in Assiut governorate. • Genetics clinic at Assiut University paediatrics' hospital., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duggan C, Irvine AD, O'B Hourihane J, Kiely ME, Murray DM. ASQ-3 and BSID-III's concurrent validity and predictive ability of cognitive outcome at 5 years. Pediatr Res. 2023 Oct;94(4):1465-1471. doi: 10.1038/s41390-023-02528-y. Epub 2023 Feb 25. PMID 36841883
- [Background] El Shafie AM, El-Gendy FM, Allahony DM, Hegran HH, Omar ZA, Samir MA, Kasemy ZA, El-Bazzar AN, Abd El-Fattah MA, Abdel Monsef AA, Kairallah AM, Raafet HM, Baza GM, Salah AG, Galab WS, Alkalash SH, Salama AA, Farag NA, Bahbah WA. Development of LMS and Z Score Growth References for Egyptian Children From Birth Up to 5 Years. Front Pediatr. 2021 Jan 18;8:598499. doi: 10.3389/fped.2020.598499. eCollection 2020. PMID 33537262
- [Background] Padeniya RN, Thushari G, Nissanka DH, Shashika C, Munasinghe DH, Aberathne DM, Weerawardena PL, Galgamuwa LS, Kumarasinghe N, Liyanage L. Maternal coping strategies in response to child's oncological diseases in Sri Lanka. Acta Oncol. 2020 Jul;59(7):866-871. doi: 10.1080/0284186X.2020.1750695. Epub 2020 Apr 14. PMID 32286131
- [Background] Waters D, Adeloye D, Woolham D, Wastnedge E, Patel S, Rudan I. Global birth prevalence and mortality from inborn errors of metabolism: a systematic analysis of the evidence. J Glob Health. 2018 Dec;8(2):021102. doi: 10.7189/jogh.08.021102. PMID 30479748
- [Background] Agana M, Frueh J, Kamboj M, Patel DR, Kanungo S. Common metabolic disorder (inborn errors of metabolism) concerns in primary care practice. Ann Transl Med. 2018 Dec;6(24):469. doi: 10.21037/atm.2018.12.34. PMID 30740400